CLINICAL TRIAL: NCT05834335
Title: Protection Against Severe Coronavirus Disease 2019 Following in Patients With Multiple Sclerosis Statified According to Disease Modifying Treatment
Brief Title: Protection Against Severe Coronavirus Disease 2019 in Patients With Multiple Sclerosis Stratified According to Disease Modifying Treatment
Acronym: PASCOMS
Status: Completed | Type: Observational
Sponsor: National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Marie D'hooghe, principal investigator, National MS Center Melsbroek
Other Study IDs: 01042023
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will conduct retrospective observational cohort study at the Nationaal Multiple Sclerose Centrum (NMSC) Melsbroek (Belgium), which is a large center specifically focusing on neurological management, multidisciplinary care and/or rehabilitation in patients with MS.

Primary endpoint For each DMT category, as defined above, the proportion of patients with a worse COVID-19 outcome (i.e., hospitalization and/or death) will be compared between those 'protected' versus 'unprotected' by vaccination at the time of SARS-CoV-2 infection. Corrections will be applied for any eventual imbalance in demographics, potentially relevant to COVID-19 outcome, between subgroups that are compared to each other, if indicated/feasible.

DETAILED DESCRIPTION:
Study design The investigators will conduct retrospective observational cohort study at the Nationaal Multiple Sclerose Centrum (NMSC) Melsbroek (Belgium), which is a large center specifically focusing on neurological management, multidisciplinary care and/or rehabilitation in patients with MS.

General aim To explore the protective effect of COVID-19 vaccination in patients with MS, stratified according to their DMT regimen (specifically isolating those treated with B-cell depleting and S1PR modulating agents), against severe forms of the infection.

Data collection Since March 2020 (i.e., the onset of the first wave of spiking COVID-19 cases in Belgium), clinical information of patients followed at the NMSC Melsbroek has been collected in a local database in case of COVID-19 diagnosis, as confirmed by positive antigen or polymerase chain reaction testing for SARS-CoV-2. The following variables were recorded: patient identification number, date of COVID-19 diagnosis, age, sex, race (White/Caucasian, Black/African-American, Asian, other), known co-morbidities (cerebro- and/or cardiovascular disease, arterial hypertension, smoking, dyslipidemia, diabetes mellitus, obesity), Expanded Disability Status Scale (EDSS) score (based on the most recent medical report prior to the infection), MS disease duration, clinical MS subtype, DMT regimen, COVID-19 severity (ambulatory care versus hospitalization versus death), general vaccination status (non-vaccinated versus fully vaccinated versus fully vaccinated + booster), date of last vaccine administration prior to the infection. On December 1, 2022, our database was locked for the present study and consisted of 450 COVID-19 cases (417 unique patients) with complete data.

Patients will be stratified according to their DMT regimen at the time of COVID-19, generating the following categories: (1) anti-CD20 B-cell depleting agents, (2) S1PR modulating agents, (3) all other forms of DMT, (4) no DMT. In each DMT category, patients will be labelled as either 'protected' or 'unprotected' by vaccination at the time of their SARS-CoV-2 infection. Patients were considered to be 'protected' by vaccination if they were (a) fully vaccinated and (b) tested positive for COVID-19 in the period ranging from 14 days to 6 months after the last administered vaccine dose (which could also be a booster).

If the DMT category at the time of last vaccination differed from that at the time of infection, patients will be excluded from the analyses; pulse corticosteroid treatment < 2 months prior to COVID-19 infection will account as an additional exclusion criterion.

Serum/plasma vitamine D levels, as measured the closest to the COVID-19 infection, if available, will be extracted from the medical record for exploratory purposes.

Primary endpoint For each DMT category, as defined above, the proportion of patients with a worse COVID-19 outcome (i.e., hospitalization and/or death) will be compared between those 'protected' versus 'unprotected' by vaccination at the time of SARS-CoV-2 infection. Corrections will be applied for any eventual imbalance in demographics, potentially relevant to COVID-19 outcome, between subgroups that are compared to each other, if indicated/feasible.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple sclerosis
* positive selftest or PCR test Coronavirus

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with multiple sclerosis and a positive selftest or positive PCR test for Corona disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
For each DMT category the proportion of patients with a worse COVID-19 outcome will be compared between those 'protected' versus 'unprotected' by vaccination at the time of SARS-CoV-2 infection. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Nationaal MS center, Melsbroek, Vlaams Brabant, Belgium